CLINICAL TRIAL: NCT02961517
Title: The Influence of Socio-demographic Characteristics on the Preferred Format of Patient Education Delivery in Individuals With Type 2 Diabetes Mellitus or Cardiovascular Disease: a Questionnaire Study
Brief Title: Format of Patient Education for Different Sociodemographic Groups
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0594
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Type2 Diabetes Mellitus; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: All patients with type 2 diabetes and/or cardiovascular disease who will complete the questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Anonymous questionnaire collecting basic sociodemographic data about the participant and information regarding their preferences for the method of delivery format of patient education information

SUMMARY:
Questionnaire study to investigate the effect of individual characteristics such as age, sex, ethnicity, educational level and socioeconomic status on the preferred format of patient education delivery, for patients with diabetes and/or cardiovascular disease

DETAILED DESCRIPTION:
An anonymous questionnaire will be used to collect basic demographic data for patients with the conditions of interest, in addition to information about their preferences for the format in which they receive patient education information. This data will be statistically analysed to address the primary and secondary outcomes of the study:

1. To investigate the effect of individual characteristics such as age, sex, ethnicity, educational level and socioeconomic status on the preferred format of patient education delivery.
2. To identify reasons for preference of patient education delivery, and whether these are associated with sociodemographic factors.
3. To assess the distribution of sociodemographic factors from participants who prefer online education, in order to identify whether preference for online education is associated with particular sociodemographic factors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over.
* Diagnosed with cardiovascular disease (defined as heart disease, peripheral vascular disease or stroke) or Type 2 diabetes
* Has not already completed the questionnaire
* Able and willing to complete questionnaire

Exclusion Criteria:

* Participant unable or unwilling to complete questionnaire
* Under the age of 18
* Not diagnosed with any of the conditions of interest
* Participant has already completed the questionnaire
* Unable to communicate (assisted or otherwise) in written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient aged 18 years or over, Diagnosed with cardiovascular disease (defined as heart disease, peripheral vascular disease or stroke) or Type 2 diabetes who has not already completed the questionnaire and is able and willing to complete questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect of sociodemographic characteristics | 9 Months
  To investigate the effect of individual characteristics such as age, sex, ethnicity, educational level and socioeconomic status on the preferred format of patient education delivery.

SECONDARY OUTCOMES:
Reasons for preferences | 9 months
  To identify reasons for preference of patient education delivery, and whether these are associated with sociodemographic factors.
Preference for online | 9 months
  To assess the distribution of sociodemographic factors from participants who prefer online education, in order to identify whether preference for online education is associated with particular sociodemographic factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Leicester Diabetes Centre, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No